CLINICAL TRIAL: NCT00778219
Title: Comparison of Autonomic Stimulation Among Different Tracheal Intubation Methods -- Using Non-invasive Heart Rate Variability Spectral Power as an Indicator
Brief Title: Comparison of Heart Rate Variability Among Tracheal Intubation Methods
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hui-Hsun Huang, visiting staff, National Taiwan University Hospital, department of anesthesiology
Other Study IDs: 200808060R
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Intubation, Endotracheal
Keywords: heart rate variability, tracheal intubation
MeSH Terms: interventions — Equipment and Supplies; Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A: Patients needing intubation of single lumen tracheal tube and performed using laryngoscope
  Interventions: Device: devices for tracheal intubation
- B: Patients needing intubation of single lumen tracheal tube and performed using lightwand
  Interventions: Device: devices for tracheal intubation
- C: Patients needing intubation of double lumen endobronchial cath and performed using laryngoscope
  Interventions: Device: devices for tracheal intubation

INTERVENTIONS:
Device: devices for tracheal intubation — tracheal intubation by laryngoscope or lightwand

SUMMARY:
60 patients, in three group of 20 patients each, scheduled for surgery needing general anesthesia will be researched. Group A: tracheal intubation of single lumen tube using laryngoscope. Group B: single lumen tube using lightwand. Group C: double lumen endobronchial cath. During general anesthesia, the spectral power of heart rate variability at three periods: (1) preoperation baseline (2) pre-intubation and (3) post-intubation will be calculated and compared to investigate the autonomic stimulation effect of different tracheal intubation methods.

DETAILED DESCRIPTION:
Tracheal intubation is a common practice during general anesthesia. Laryngoscope and lightwand are two commonly used methods of tracheal intubation. The autonomic stimulation of tracheal intubation may have adverse effect to the patients and have been investigated since many years ago. Conventional methods for assessing autonomic activity include measurement of blood catecholamine levels or measuring changes of the hemodynamic variables such as heart rate and blood pressure. The former is invasive and noncontinuous, and the latter is nonspecific and not accurate. Heart rate variability, a parameter derived from the spectral power of RR interval sequence in the ECG, is a non-invasive but direct measurement of autonomic activity. It is ideal and we will use this in the current research for comparing the autonomic activation during tracheal intubation of the two different methods.

Totally 60 ASA class I-II patients aged 18-65 years will be recruited. 40 of these are scheduled for various kind of surgery needing general anesthesia with tracheal intubation of single lumen tube. These 40 patients will be randomly assigned into group A and B, each with 20 patients. In group A the tracheal intubation will be performed by laryngoscope, and in group B the intubation performed by lightwand. The other 20 patients of the study, the group C, are scheduled for operations needing intubation of double lumen endobronchial cath. The intubation will be performed by laryngoscope.

ECG wil be recorded from at least 5 minutes before induction of general anesthesia and continue to at least 10 minutes after tracheal intubation. The induction and maintenance of anesthesia will performed as routine practice. The ECG records wil be analyzed offline. Power spectrum wil be generated by time-frequency analysis and the heart rate variability parameters at three periods (1)preoperation baseline (2) pre-intubation and (3) immediately post-intubation will be calculated and compared among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-II, age 18-65, scheduled for surgery needing general anesthesia with tracheal intubation

Exclusion Criteria:

* history of major systemic diseases such as cardiovascular, pulmonary, renal and other diseases which affect autonomic activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 ASA class I-II patients , age 18-65, scheduled for surgery and need general anesthesia with tracheal intubation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
spectral power of heart rate variability | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsun Huang, MD, PhD, Principal Investigator — Department of anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan